CLINICAL TRIAL: NCT03890549
Title: Validation of Downloadable Mobile Snore Applications by Polysomnography
Brief Title: Validation of Downloadable Mobile Snore Applications by Polysomnography (PSG)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201801799B0
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-12

CONDITIONS: Apnea, Obstructive; Snoring
Keywords: obstructive sleep apnea; polysomnography; smart phone application
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obstructive sleep apnea group: The patients were diagnosed by thoracic and ENT (Eye-Nose-Throat) specialist through polysomnography.
  Interventions: Diagnostic Test: SnoreLab (smart phone application for snoring recording)

INTERVENTIONS:
Diagnostic Test: SnoreLab (smart phone application for snoring recording) — The investigators selected 3 appropriate downloadable smart phone applications for snoring recording and make validation with the golden standard of polysomnography.
  Other Names: Sleep Cycle alarm clock (smart phone application for snoring recording); Anti Snore Solution (smart phone application for snoring recording)

SUMMARY:
The aim of this study is to validate the downloadable mobile snore applications by polysomnography.

DETAILED DESCRIPTION:
Obstructive sleep apnea(OSA) is characterized by multiple episodes of upper airway collapse during sleep and considered as a major health issue worldwide due to comorbidity with obesity, hypertension, diabetes and more advanced cardiovascular diseases. The noisy sounds of snoring caused by OSA bother bed partner sleepless and lead to long-term health problems. Mobile snore applications are convenient and accessible for patients to monitor the progress of OSA by themselves, but there are no reliable PSG-validated applications.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign inform consent with aged more than 20 years old
* Mild to moderate OSA, AHI (apnea-hypopnea index) < 30

Exclusion Criteria:

* Significant lung disease
* Skeletal facial framework problems
* Central apnea
* Receiving acupuncture in recent 2 weeks
* Taking hypnotic drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed as obstructive sleep apnea no matter disease severity.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
snore time | through study completion during sleep, each sleep cycle about 6-8 hours
  snoring time during sleep accessed by PSG and smart phone applications
snore counts | through study completion during sleep, each sleep cycle about 6-8 hours
  snoring counts during sleep accessed by PSG and smart phone applications
snore sound | through study completion during sleep, each sleep cycle about 6-8 hours
  snoring sound during sleep accessed by PSG and smart phone applications
sleep time | through study completion during sleep, each sleep cycle about 6-8 hours
  total sleep time accessed by PSG and smart phone applications

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No
1. There will be a research number representing the identity. This number will not display the name, identification number, and address.
  2. For the results and diagnosis of the visit, the research host will maintain a confidential attitude and carefully maintain the privacy. If research results are published, the identity will remain confidential.
  3. Please also understand that if the participant signs the consent form, the participant agrees that the visit record can be directly reviewed by the monitor, auditor, research ethics committee and the competent authority to ensure that the research process and data comply with relevant laws and regulations. These people also promise not to violate the confidentiality of your identity.